CLINICAL TRIAL: NCT02500810
Title: A Randomized, Controlled, Multicenter Phase II Clinical Trial of Monosialoganglioside(GM1) Preventing Neurotoxicity Induced by Albumin-bound Paclitaxel Chemotherapy in Lung Cancer Patients
Brief Title: Monosialoganglioside Preventing Neurotoxicity Induced by Albumin-bound Paclitaxel Chemotherapy in Lung Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Peking University First Hospital (Other); Peking University Third Hospital (Other); Chinese PLA General Hospital (Other); Peking Union Medical College Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Beijing Shijitan Hospital, Capital Medical University (Other); Yantai Yuhuangding Hospital (Other); Weifang People's Hospital (Other)
Responsible Party: Principal Investigator, Jian Fang, Director of Thoracic Onconlogy Department, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GW-N-1501
Record Dates: First submitted 2015-07-11; First posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Neurotoxicity
Keywords: neurotoxicity; chemotherapy; monosialoganglioside; prevention
MeSH Terms: conditions — Neurotoxicity Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- monosialoganglioside (Experimental): patients receive monosialoganglioside.
  Interventions: Drug: monosialoganglioside
- control (No Intervention): blank control

INTERVENTIONS:
Drug: monosialoganglioside — 40mg in the vein on day 1 - day 8 of each 21 days cycle. Number of Cycles: 2 cycles.
  Other Names: GM1; Monosialotetrahexosylganglioside Sodium Injection
  Arms: monosialoganglioside

SUMMARY:
The purpose of this study is to determine whether monosialoganglioside are effective in the prevention of neurotoxicity induced by albumin-bound paclitaxel chemotherapy in lung cancer patients, and improve the quality of life of patients.

DETAILED DESCRIPTION:
Lung cancer patients received a single-agent albumin-bound paclitaxel chemotherapy are included in this trial. Patients are randomly assigned into the experimental group and blank control group based on segmented block randomized method. After enrollment, patients will complete at least chemotherapy and GM1 injection/blank control. During the 3w per cycle chemotherapy, albumin-bound paclitaxel is conducted in D1 and D8, GM1(40mg+250ml N.S) is injected from D1 to D8. Neurotoxicity evaluation and quality of life assessment will be conducted every cycle and 3m/6m after the chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Cytological and histological confirmation of unresectable locally advanced or metastatic lung cancer diagnosis
* No peripheral nervous system diseases exists before
* Within 4 weeks before treatment, did not receive other adverse reaction of drugs may cause similar neurotoxicity
* Enough organ functions reservation and appropriate performance status for chemotherapy
* Expected survival period is more than 3 months

Exclusion Criteria:

* Known or assignment of any of these products to test drugs allergic agent composition
* With peripheral neuropathy by any cause before treatment
* With other neurological dysfunction which can cause inaccurate record of the occurrence of neurotoxicity and severity
* Patients with poor general condition to receive chemotherapy
* Genetic glucolipid metabolic abnormalities
* Patients (male or female) have fertility possibility but not willing to or not to adopt effective contraception
* Patients cann't avoid neurotrophic drugs
* According to the researcher's judgment, the situations inappropriate for patients with ganglioside medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
incidence of neurotoxicity | up to 4 weeks after the 2nd cycle albumin-bound paclitaxel chemotherapy

SECONDARY OUTCOMES:
time(days）neurotoxicity arise | up to 6 months neurotoxicity after the first use of albumin-bound paclitaxel chemotherapy
Peripheral nerve conduction velocity | up to 4 weeks after the albumin-bound paclitaxel chemotherapy

OTHER OUTCOMES:
time(days) of neurotoxicity adverse events alleviation | up to 180 days after the albumin-bound paclitaxel chemotherapy
quality of life | up to 4 weeks after the albumin-bound paclitaxel chemotherapy
side effects of monosialoganglioside | up to 4 weeks after the albumin-bound paclitaxel chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jian Fang, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China